CLINICAL TRIAL: NCT07321275
Title: Ultra-early Chest CT Improves Risk Prediction of Stroke-associated Pneumonia: Model Development and External Validation in a Multicentre Retrospective Study
Brief Title: Ultra-early Chest CT for SAP Prediction
Acronym: SENTRY
Status: Recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor of Neurology, Xuanwu Hospital, Capital Medical University, Capital Medical University
Other Study IDs: SENTRY
Record Dates: First submitted 2025-12-19; First posted 2026-01-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischaemic Stroke; Stroke-associated Pneumonia
Keywords: Acute ischaemic stroke; Stroke-associated pneumonia; Risk prediction model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Development (Derivation) cohort
- External validation cohort

SUMMARY:
Stroke-associated pneumonia (SAP) is a common and serious complication after acute ischaemic stroke (AIS). Existing scores rely mainly on clinical variables, and the added prognostic value of inflammatory markers and early chest CT findings remains uncertain. We developed and externally validated an early multimodal model combining clinical severity, inflammation, and chest CT abnormalities, and explored risk-stratified associations between prophylactic antibiotics and SAP.

ELIGIBILITY:
Inclusion criteria:

1. patients aged ≥18 years;
2. Admitted to a participating stroke centre with neuroimaging-confirmed acute ischaemic stroke ;
3. Had chest CT performed within 24 hours of stroke onset.

Exclusion criteria:

1. Pneumonia;
2. Chest CT images unavailable or incomplete for assessment;
3. Insufficient clinical documentation to ascertain stroke-associated pneumonia occurrence within 7 days after stroke onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with neuroimaging-confirmed acute ischemic stroke admitted to participating tertiary stroke centers in China. Eligibility requires chest CT performed within 24 h of stroke onset . Patients will be retrospectively identified from electronic medical records and stroke registries, and stroke-associated pneumonia will be assessed within 7 days after stroke onset using prespecified criteria. Only the first eligible admission per individual will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Stroke-associated pneumonia | within 7 days after stroke onset
  SAP was defined as pneumonia occurring within 7 days after stroke onset. Potential events were screened using discharge diagnosis codes and medical record documentation, and then confirmed by manual chart review using prespecified clinical, laboratory, and radiological criteria consistent with the Pneumonia in Stroke Consensus Group and modified CDC definitions.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Suzhou Municipal Hospital of Anhui Province, Suzhou, Anhui
  - Rongcheng County People's Hospital, Baoding, Hebei
  - Ningjin County People's Hospital, Fenghuang, Hebei
  - The Second Hospital of Hebei Medical University,, Shijiazhuang, Hebei
  - Central Hospital of Xiangtan, Xiangtan, Hunan
  - First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Shihezi People's Hospital,, Shihezi, Xinjiang
  - Xuanwu Hospita, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Related data will be shared if full study protocol and statistical analysis plan are provided with reasonable design.